CLINICAL TRIAL: NCT07156526
Title: Safety and Efficacy of Two Qualia Iron Formulations on Iron Biomarkers and Quality of Life: A Randomized, Double-Blind Pilot Study
Brief Title: Impact of Two Iron Formulations on Iron Biomarkers and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: QLS-015
Record Dates: First submitted 2025-08-12; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Iron Deficiencies
Keywords: Iron supplementation; Iron deficiency
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qualia Iron Version A (Active Comparator): Qualia Iron version A manufactured by Qualia Life Sciences
  Interventions: Dietary Supplement: Qualia Iron Version A
- Qualia Iron Version B (Active Comparator): Qualia Iron version B manufactured by Qualia Life Sciences
  Interventions: Dietary Supplement: Qualia Iron Version B
- Placebo (Placebo Comparator): Rice powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia Iron Version A — Qualia Iron Version A manufactured by Qualia Life Sciences
  Arms: Qualia Iron Version A
Dietary Supplement: Qualia Iron Version B — Qualia Iron Version B manufactured by Qualia Life Sciences
  Arms: Qualia Iron Version B
Dietary Supplement: Placebo — Rice powder
  Arms: Placebo

SUMMARY:
This randomized, double-blind parallel pilot study will evaluate the safety and efficacy of two Qualia Iron formulations versus placebo in approximately 40 healthy adults (aged 18+) over a 56-day period. Approximately 40 participants will be randomized to three study arms: Qualia Iron Version 1, 2, (n=15 each) or a Placebo (n=10). Each participant will take one or two capsules once daily in the morning, with or without food. The supplementation regimen is a 5 days on, 2 days off protocol, and goes for 56 days (8 weeks). The primary outcomes of this study are to assess between-group changes in iron status biomarkers. Secondary outcomes include within-group changes in iron status biomarkers, safety and tolerability as measured by a custom Safety and Tolerability survey, and RAND SF-36 quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary, written, informed consent to participate in the study
* Agree to provide a valid cell phone number and are willing to receive communications through text
* Can read and write English
* Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly
* Willing to complete questionnaires, records, and diaries associated with the study.
* If the participant responded "Yes" to ≥2 questions on the custom Iron Inadequacy Questionnaire. Preference will be given to participants with a higher score.
* If a participant has the following:

Ferritin 30 ng/mL (anything under 50 ng/mL is considered suboptimal, but participants with 30 ng/mL will be prioritized)

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
* Known food intolerances/allergy to any ingredients in the product
* Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, irritable bowel disease, cancer
* Having had a significant cardiovascular event in the past 6 months
* Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines
* On immunosuppressive therapy
* Individuals who were deemed incompatible with the test protocol
* Adults lacking capacity to consent
* Individuals taking any of the following medications:

Antacids Proton pump inhibitors (PPIs) Antipsychotics Antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Changes in iron status biomarkers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Between-groups changes in ferritin levels (ng/mL) will be assessed.

SECONDARY OUTCOMES:
Changes in iron status biomarkers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in serum iron (mcg/dL)
Changes in iron status biomarkers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in percent saturation (%)
Changes in iron status biomarkers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in total iron binding capacity (mcg/dL)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in hematocrit (%)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in hemoglobin (g/dL)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in red cell distribution width (%)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in mean corpuscular volume (fL)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in mean corpuscular hemoglobin (pg)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in mean corpuscular hemoglobin concentration (g/dL)
Changes in CBC markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in red blood cell count (million/microliter)
Changes in RAND 36-Item Short Form Survey (SF-36) | From 0-4 weeks, 4-8 weeks, 0-8 weeks
  The RAND SF-36 captures 8 separate aspects of health-related quality of life using the same 0-to-100 scoring scale for all eight domains. Higher scores represent better health outcomes.
Changes in Safety and Tolerability measured by Custom Survey | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in safety and tolerability measures will be examined in each group using a custom survey. The survey asks about common nocibo side effects, including increasing anxiety/worry, headache, mood changes, stomach upset/nausea, dizziness, bloating, itching, and sexual function. The scoring system goes from "not at all" to "a great deal" for each item, . The total score for each category across all participants will be calculated, and then timepoint comparisons will be made.
Changes in inflammatory markers | From 0-4 weeks, 4-8 weeks, and 0-8 weeks
  Changes in high sensitivity C-reactive protein (mg/L)
Changes in iron status biomarkers | From 0-4 weeks, 4-8 weeks and 0-8 weeks
  Within-groups changes in ferritin (ng/mL) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: William Scuba, Principal Investigator — Qualia Life Sciences
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No